CLINICAL TRIAL: NCT06866145
Title: Dexmedetomidine Infusion in Either Total Intravenous Anesthesia or Inhalational Anesthesia to Improve Surgical Field Visibility in Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3/2024 ANE T8
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-03

CONDITIONS: Rhinosinusitis
Keywords: endoscopic sinus surgery , dexmedetomidine, surgical field visibility
MeSH Terms: conditions — Rhinosinusitis | interventions — Dexmedetomidine

STUDY DESIGN:
Masking Description: surgeon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TIVA group (Other): patients receives total intravenous anesthesia
  Interventions: Procedure: functional endoscopic sinus surgery; Drug: Dexmedetomidine
- inhalational group (Other): patients receives inhalational anesthesia
  Interventions: Procedure: functional endoscopic sinus surgery; Drug: Dexmedetomidine

INTERVENTIONS:
Procedure: functional endoscopic sinus surgery — sinus surgery
Drug: Dexmedetomidine — precedex

SUMMARY:
Dexmedetomidine Infusion in either Total Intravenous Anesthesia or Inhalational Anesthesia to Improve Surgical Field Visibility in Endoscopic Sinus Surgery

DETAILED DESCRIPTION:
the study was prospective randomized single blinded study

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I and II patients undergoing endoscopic sinus surgery in the age group from 18-50 years.

Exclusion Criteria:

* History of allergy to medications used in the study, refusal of patients to participate, hepatic or renal dysfunction, chronic pain condition, psychological and neurological disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Surgical field visibility | intraoperative
  Surgical field visibility assessed every 15 minutes based on Boezaart scale from 0 to 5 as 0 is the worst score and 5 is the best

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Menoufia university hospital, Menoufia, Shibin Elkom
  - Menoufia university hospital, Shibin Elkom